CLINICAL TRIAL: NCT04886219
Title: Studies of the Characteristics of the Angle Kappa and the Angle Alpha in the Healthy Individual. Studies of the Angle Kappa and the Angle Alpha
Brief Title: Studies of the Angle Kappa and the Angle Alpha
Acronym: EKAPS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210289; 2020-A03370-39 (Other: IDRCB number)
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: No Eye Disorder
Keywords: Angle Kappa; Angle Alpha; Pupillary axis; Visual axis; Optical axis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy individual: Healthy individual
  Interventions: Other: Eye examination

INTERVENTIONS:
Other: Eye examination — * Multimodal fundus imaging (color fundus photography, optical coherence tomography (OCT))
  * orthoptic assessment (Visual acuity, Refraction, Cover test, Stereopsis evaluation
  * ocular biometry
  * corneal topography
  * monocular photographs in photopic and scotopic condition

SUMMARY:
Anatomical ophthalmological connections and their dynamics are still debated in the scientific community. However, their considering is essential in many surgeries (strabismus, cataract, refractive...) or in clinical practice.

The correlation between these biometric values would make it possible to refine the knowledge related to these landmarks and thus offer better ophthalmological management by integrating these variables into the clinical examination.

The aim of the study is to analyze the correlation between the angle alpha and the angle kappa in a healthy individual without ophthalmologic disorder.

DETAILED DESCRIPTION:
The angle kappa corresponds to the angle formed between the visual axis (line between the point of fixation and the fovea: area of the retina allowing precise vision) and the pupillary axis (line passing through the center of the pupil and perpendicular to the cornea). The angle alpha corresponds to the angle formed between the visual axis and the optical axis (line passing through the nodal point of the eye and corneal center).

In theory, the angle kappa and angle alpha are equal; but physiological corectopy in the nasal position induces a variation between these two angles; the angle kappa being generally less than the angle alpha without a correlation being established. Also, pupillary constriction causes a variation in the position of the center of the pupil. The angle kappa therefore exhibits a variation depending on the expansion.

Anatomical ophthalmological connections and their dynamics are still debated in the scientific community. However, their considering is essential in many surgeries (strabismus, cataract, refractive ...) or in clinical practice.

The correlation between these biometric values would make it possible to refine the knowledge related to these landmarks and thus offer better ophthalmological management by integrating these variables into the clinical examination.

The aim of the study is to analyze the correlation between the angle alpha and the angle kappa in a healthy individual without an eye disorder.

ELIGIBILITY:
Inclusion Criteria:

- Informed major subject not opposing to their participation in the study

Exclusion Criteria:

- Subject with strabismus or organic ophthalmologic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy individuals without visual disorders
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Value of the angle Kappa | Day 0
  Semi-automatic digital method of measurement by eye photography
Value of the angle Alpha | Day 0
  Semi-automatic digital method of measurement by eye photography

SECONDARY OUTCOMES:
Variation of the Kappa angle depending on the pupillary diameter | Day 0
  Variation in the same individual. Value of the Kappa angle using the semi-automatic method of measurement by ocular photography in photopic and scotopic conditions & measurement of the pupillary diameter using the photographs obtained
Correlation between the value of the angle Alpha and the Optic disc / fovea distance | Day 0
  Angle Alpha value using the semi-automatic method of measurement by eye photography and the distance between the optic disc and the fovea
Correlation between the angle Kappa and the axial length | Day 0
  Value of the angle Kappa and Alpha using the semi-automatic method of measurement by eye photography and Value of the axial length measured by biometry IolMaster 500 (Carl Zeiss)

CONTACTS AND LOCATIONS:
Overall Officials: Maxence Rateaux, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique Brémond-Gignac, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rateaux M, Vienne-Jumeau A, Bremond-Gignac D, Robert MP. Fluctuations in angle lambda with the pupil diameter and correlations with biometric values in a healthy population. Ophthalmic Physiol Opt. 2025 Nov;45(7):1837-1844. doi: 10.1111/opo.70006. Epub 2025 Aug 14. PMID 40810703
- [Background] Rateaux M, Bremond-Gignac D, Robert MP. From monocular photograph to angle lambda: A new clinical approach for quantitative assessment. J Binocul Vis Ocul Motil. 2022 Jul-Sep;72(3):169-175. Epub 2022 Jun 22. PMID 35731900